CLINICAL TRIAL: NCT04842110
Title: A Prospective, Controlled, Standardized, Multi-center, Single-treatment, Single- Arm Evaluation of the EonTM FR 1064 nm Device to Reduce Abdominal Fat
Brief Title: Eon™ FR 1064 Full Abdomen Clinical Study Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dominion Aesthetic Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D0000000151
Record Dates: First submitted 2021-04-08; First posted 2021-04-13 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Abdominal Obesity
MeSH Terms: conditions — Obesity, Abdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- 1064 Full Abdomen (Experimental): eonTM FR 1064 nm device Patient will be treated with the eonTM FR 1064 nm device
  Interventions: Device: Experimental: eonTM FR 1064 nm device

INTERVENTIONS:
Device: Experimental: eonTM FR 1064 nm device — The subject treatment area - abdomen, was treated with the 1064 nm wavelength laser.

SUMMARY:
This is a marketing study intended to provide additional data for marketing purposes for the eon™ FR is FDA 510(k) which has been cleared for non-invasive lipolysis of the abdomen to achieve disruption of adipocyte cells intended for non-invasive aesthetic use to achieve a desired aesthetic effect. This device is intended for individuals with a Body Mass Index (BMI) of 30 kg/m2 or less.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a healthy male or female > 18 years or older seeking treatment for unwanted fat in the abdomen.
* Subject must be able to read, understand and sign the Informed Consent Form (ICF) in English.
* Subject has sufficient thickness (≥ 25 mm) of adipose tissue on the abdomen area.
* Study subjects must agree to maintain their current diet and weight (not gaining or losing greater than ±5 lbs.
* Subject must be willing and able to adhere to the treatment and follow-up visit schedule.
* Subject must be willing to have limited sun exposure for the duration of the study, including the follow-up period.
* Subject is willing to have photographs and ultrasound measurements taken of the treated area, which will be de-identified in evaluations and may be used in presentations and/or publications.
* Female subjects must be using medically acceptable form of birth control during the entire course of the study or may be post-menopausal, surgically sterilized.

Exclusion Criteria:

* Aesthetic fat reduction procedure in the treatment area within the previous year.
* Pregnant in the last 3 months, intending to become pregnant, postpartum or nursing in last 6 months
* Unstable weight within the last 6 months (+ or - 3% weight change in the prior six months)
* Subject has an infection, dermatitis or a rash in the treatment area.
* Subject has tattoos or jewelry in the treatment area or within the treatment area site or photography frame.
* Subject has a history of keloid scarring, hypertrophic scarring or of abnormal wound healing.
* Subject has a history of immunosuppression/immune deficiency disorders or currently using immunosuppressive medications.
* Subject has a history of a known bleeding disorder.
* Subject has a known photosensitivity to the study laser wavelength, history of ingesting medications known to induce photosensitivity, or history of seizure disorders due to light.
* Subject has known collagen, vascular disease or scleroderma.
* Subject has undergone a surgery or procedure in the treatment area within 6 months of treatment, which is still healing.
* Subject suffers from significant concurrent illness, such as insulin-dependent diabetes, peripheral vascular disease or peripheral neuropathy.
* Subject is undergoing systemic chemotherapy for the treatment of cancer.
* Subject is using gold therapy for disorders such as rheumatologic disease or lupus.
* Subject has participated in a study of another device or drug within three months prior to enrollment or during the study.
* As per the investigator's discretion, the subject has any physical or mental condition which might make it unsafe for the subject to participate in this study.
* Subject has ongoing use of steroids or secondary rheumatoid drugs.
* Subject is actively taking psychotropic medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-08-24 (Actual); Primary Completion 2019-12-21 (Actual); Study Completion 2019-12-21 (Actual)

PRIMARY OUTCOMES:
Photographic Evaluations as a Measure of Effectiveness | 12 Weeks
  Photographs of the treatment area will be obtained at baseline and 12 weeks post treatment and be evaluated by blinded independent readers to correctly identify pre-treatment (baseline) photographs compared to 12 weeks post treatment photographs in order to determine effectiveness of device.

SECONDARY OUTCOMES:
Change in Adipose Layer Thickness | 12 weeks
  Ultrasound measurements of adipose layer thickness will be collected at baseline and 12 weeks after procedure to evaluate changes between both.
Subject Satisfaction | 12 weeks
  Subject Questionnaires will be completed by subjects at the end of study to determine the subject satisfaction with procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Fiala Aesthetics, Altamonte Springs, Florida, United States

IPD SHARING:
Plan to Share IPD: No